CLINICAL TRIAL: NCT02039310
Title: Prediction of Impaired Survival in Elderly Bladder Cancer Patients Opting for Radical Cystectomy
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Cheryl Lee, PI, University of Michigan
Other Study IDs: HUM00057382
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine, serum, psoas muscle specimen

GROUPS / COHORTS (1):
- ≥ 65 years / opts for radical cystectomy

SUMMARY:
The investigators proposes a prospective cohort study in patients with high risk bladder cancer who have opted for radical cystectomy. The investigators aim to correlate pre-operative measures of body composition, cognitive and functional status with impaired survival at 6 months after cystectomy. Impairment in this context will be a compilation of several specific objective measures including: 1) death from any cause, 2) major complication (Clavien score7 ≥ 3), 3) loss of independent living status, 4) performance status, and 5) global well-being. The study team believes that Impairment Free Survival is an important endpoint as it accounts for many aspects of a patient's functional status that might alter a patient's choice to proceed with radical surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of bladder carcinoma (any histology permitted)
* Planned treatment with radical cystectomy.
* Age 65 years or older at the time of radical cystectomy
* Able to give consent
* Neoadjuvant chemotherapy is permissible
* Prior malignancy is permissible, without evidence of disease for at least 2 years
* Concomitant localized prostate cancer, skin cancer, and in situ malignancies are permissible.
* Willingness to complete surgical follow-up at the University of Michigan for at least 6 months after radical cystectomy.

Exclusion Criteria:

* Evidence of metastatic bladder cancer
* Life expectancy less than one year
* Concurrent treatment on another clinical trial. Non-intervention supportive care trials or non-treatment trials, e.g. QOL, are allowed

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients meeting eligibility criteria will be recruited from genitourinary cancer clinics at the University of Michigan Comprehensive Cancer Center. Patients undergoing initial consultation, active treatment, or surveillance after endoscopic or intravesical therapy will be identified and screened. Interested patients will be counseled by Dr. Lee or her designee, who will review the rationale and benefits of the study, the potential risks and probability of their occurrence, and the procedures to minimize these risks. Patients who wish to enter the study will be asked to sign a consent form that meets the requirements of the University of Michigan IRB. A signed copy of the patient consent will be entered into the medical record.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Impairment Free Survival | 6 months
  Impairment-free survival is defined as the time from radical cystectomy to the identification of: 1) major complication (Clavien score7 ≥ 3), 2) loss of independent living status, 3) ECOG performance status ≥ 3 beyond 4 weeks from RC, 4) global well-being or 5) death from any cause. Patients who drop-out before the 6-month end of study and who have not had an impairment event will be censored at their time of drop-out.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl T Lee, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States